CLINICAL TRIAL: NCT04997707
Title: The Effect of Propofol-based Anaesthesia Versus Low Dose Propofol With Less Than Half MAC Sevoflurane on Intraoperative Trans-cranial Motor Evoked Potential During Spine Surgeries: Ratios Rather Than Values.
Brief Title: The Effect of Balanced Anesthesia Regimen on Intraoperative Trans-cranial Motor Evoked Potential During Spine Surgeries:
Acronym: NIOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: El-Sahel Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Samir Ahmed Ahmed ElKafrawy, consultant of anesthesia, head of neuroanesthesia unit, El-Sahel Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 322018
Record Dates: First submitted 2021-07-14; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Motor Evoked Potential
Keywords: motor-evoked potentials, sevoflurane, balanced anesthesia,
MeSH Terms: interventions — Propofol; Sevoflurane; Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P group (Active Comparator): 75-100 µg/kg/min propofol
  Interventions: Drug: Propofol Abbott; Diagnostic Test: transcranial motor evoked potential(Tcm
- BA group (Active Comparator): 25ug/kg/min propofol and 0.2% below corrected-to-age- half MAC of sevoflurane
  Interventions: Drug: Propofol Abbott; Drug: Sevoflurane Inhalation Solution; Diagnostic Test: transcranial motor evoked potential(Tcm

INTERVENTIONS:
Drug: Propofol Abbott — in a rate of 75-100 μg/kg/min in P group, and 25μg/kg/min in BA group
  Other Names: propofol
Drug: Sevoflurane Inhalation Solution — in BA group will be calculated by age-adjusted end - tidal MAC as follows: for age of 18-25 years, 26-40 years and ≥40 years MAC will be 2.6%, 2.2% and 1.8% respectively then final concentration to be delivered will be 0.2% lower than calculated half MAC.
  Other Names: sevoflurane
  Arms: BA group
Diagnostic Test: transcranial motor evoked potential(Tcm — using NIM-SPINE™ SYSTEM (2005 Medtronic Sofamor Danek USA, Inc.). The stimulation used is a train-of-five square wave stimulation, 2ms inter-stimulus interval, 500 μs width and 40-220 mA intensity which can be increased with 10 mA steps till muscle answer potential is recorded.
  Other Names: intraoperative neurophysiological monitoring (IONM)

SUMMARY:
transcranial motor evoked potentials (TcMEP) were proved to be useful during complicated spinal surgeries to prevent iatrogenic complications. The effect of anesthetic agents was comprehensively discussed in literature. The Investigators studied a new balanced anesthetic protocol using propofol and sevoflurane in addition to continuous fentanyl infusion in which they compared values and ratios of amplitudes and latencies of TcMEP waves at different time point.

DETAILED DESCRIPTION:
This is a prospective double- blind randomized controlled study. After approval by the ethics committee at the National Cancer Institute (Cairo University) and El-Sahel Teaching Hospital (GOHTI, Cairo) and after written informed consents,46 ASA I-II patients who are scheduled for various spinal surgeries (such as: intra-spinal tumor resection, spondylolisthesis correction, traumatic spinal fractures' fixation,…) will be included in this study. Surgeons and neurophysiologists will be the same and will be blind to the anesthetic techniques in all patients.

Randomization list will be generated then patients will be randomized into two groups: control and study group.

Preoperatively, all patients will be checked for any exclusion criteria and the routine preoperative evaluation will be done. On arriving operative theater, all patients will receive 0.1 mg/kg midazolam IV. After connecting all the basic monitors' cables (NIBP, pulse oximetry and ECG) and canulating the radial artery to monitor IBP, induction of anesthesia will be done to all patients with 4μg/kg fentanyl, 2-3mg/kg propofol IV and 0.5mg/kg atracurium to facilitate endotracheal intubation. After intubation, central venous catheter( CVP), temperature probe through nasopharynx and urinary catheter will be inserted. Fentanyl infusion will be maintained in a rate of 2μg/kg/hour and will be discontinued 60 minutes before recovery.

From this time on, patients will be randomly allocated into control and study groups, each group is 30 patients; control group is the propofol (P) group and the study group is the balanced anesthesia (BA) group.

Control Group: propofol will be infused continuously in a rate of 75-100 μg/kg/min Study Group: propofol infusion in a rate of 25μg/kg/min will be given with sevoflurane. Sevoflurane concentration will be individually calculated by age-adjusted end - tidal MAC as follows: for age of 18-25 years, 26-40 years and ≥40 years MAC will be 2.6%, 2.2% and 1.8% respectively then final concentration to be delivered will be 0.2% lower than calculated half MAC.

Patients will be mechanically ventilated with O2/Air mixture (FiO2 50%) in a rate of 10-12/minute and tidal volume of 6-8 ml/kg to insure oxygen saturation (SpO2) around 99% and end-tidal CO2 between 28-35 mmHg. Body temperature must be kept between 35-37oC( Celsius degrees) using warm fluids and warming blankets.

Intraoperative fluids will be given guided by central venous pressure (CVP)and urine output.

Hypotension ( mean arterial blood pressure (MAP) ˂60 mmHg in normotensive patients or ˂70 mmHg in hypertensive patients) will be treated with Norepinephrine (Levophed®) in an infusion of 0.05-1.0μg /kg/min.

TcMEP Monitoring:

After induction, transcranial stimulation electrode will be connected at C1- C2, Cz and C3-C4 (10-10 international system) and subdermal needles inserted in the appropriate muscles, according to the scenario selected, processing will be done using NIM-SPINE™ SYSTEM (2005 Medtronic Sofamor Danek USA, Inc.). The stimulation used is a train-of-five square wave stimulation, 2ms inter-stimulus interval, 500 μs width and 40-220 mA intensity which can be increased with 10 mA steps till muscle answer potential is recorded.

The first TcMEP (R1) will be taken before positioning and surgical incision, at least 20-25 minutes after induction; fading of the neuromuscular blockade will be checked by train-of-four (TOF) and double- burst stimulation using peripheral nerve stimulator connected to the ulnar nerve.

A second reading (R2), which is the surgical baseline reading, will be taken 20 minutes later; during which positioning of the patient is done; again muscle relaxant fading is confirmed before the reading as above. A third reading (R3) will be taken after the surgical incision.

With every TcMEP reading, MAP, pulse rate, Oximetry, En-tidal CO2, nasopharyngeal temperature, ulnar train-of-four response, sevoflurane percentage concentration / propofol infusion rate and CVP will be recorded.

Comparison between R1 and R2 will be dedicated to the effect of anesthetic regimen, while subsequent readings will indicate both the effect of anesthetic regimen and any surgical insult (if any).

Decrease in every wave amplitude by more than 50% in relation to R1 and increase in latency more than 2 ms will be recorded as an alarming criterion.

On recovery:

After fulfilling the Modified Aldrete Recovery Score, patients will be discharged from postoperative recovery unit (PACU) to the intermediate care unit. All patients with an alarming criterion will be checked by neurosurgeon for any motor deficit.

Sample size estimation:

The aim of this study is to compare the effects of balanced anesthesia using low dose propofol and less than half MAC sevoflurane versus propofol based anesthesia while using medium-dose fentanyl in both techniques on TcMEP intraoperative monitoring during spine surgeries. Based on the previous paper published by Palazon et al., 2015, the difference in latency between the 2 groups was 3 with an average variability of 3. A total sample size of 46 (23 per group) will be sufficient to detect that effect size, with power 90% and 5% significance level the sample size was calculated by the G power program.

ELIGIBILITY:
Inclusion Criteria:

* (ASA) grades I-II who were scheduled for spinal surgeries (intraspinal tumors resection, spondylolisthesis correction, traumatic spinal fractures fixation….etc)

Exclusion Criteria:

* Patients aged less than 18 years, or with history of drug abuse, any pulmonary disease, preoperative motor deficit, history of epilepsy, pacemakers and cochlear implants, previous intracranial surgeries or needed to deepen anesthetic plane during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — More than 18 years
Enrollment: 60 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
TcMEP Monitoring (R1) | " up to 45 minutes"
  The first TcMEP (R1) was taken before positioning and surgical incision, at least 20-25 min
TcMEP Monitoring(R2) | "up to 60 minutes"
  R2), after positioning of the patient
TcMEP Monitoring(R3) | " up to 75 minutes"
  (R3) was taken after the surgical incision

SECONDARY OUTCOMES:
Mean arterial blood pressure (MAP) | " up to 5 hours"
  in mmHg
pulse rate | " up to 5 hours"
  number / minute
Spo2 | " up to 5 hours"
  in percentage
temperature | " up to 5 hours"
  in C
propofol infusion rate | " up to 5 hours"
  ml/hour
end-tidal sevoflurane | " up to 5 hours"
  percentage
Central venous pressure (CVP) | " up to 5 hours"
  cmH2O
end-tidal CO2 | " up to 5 hours"
  mmHg
PaO2 | " up to 5 hours"
  mmHg
PaCo2 | " up to 5 hours"
  mmHg
PHa | " up to 5 hours"
  Number
Train-of-four stimulation ( TOF) | " up to 5 hours"
  percentage
R3/R2 ratio | " up to 5 hours"
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Samir A El kafrawy, MD, Principal Investigator — El-Sahel Teaching Hospital
Locations (2):
- Egypt (2):
  - National cancer Institute, Cairo
  - El sahel Teaching Hospital, Cairo

IPD SHARING:
Plan to Share IPD: No
Methods and results